CLINICAL TRIAL: NCT01303211
Title: A Case-control Study of the Efficacy of a New Serogroup A Meningococcal Conjugate Vaccine (MenAfriVac) in Mali and Niger
Acronym: VES
Status: Withdrawn | Type: Observational
Why Stopped: No cases on NmA meningitis were recorded following vaccination with MenAfriVac
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: VES_5840
Record Dates: First submitted 2011-02-08; First posted 2011-02-24 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal serogroup A conjugate vaccine; Vaccine efficacy; Serogroup A meningococcal diseases
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sera samples will be separated from 5 ml blood sample obtained from cases and controls.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- serogroup A meningococcal disease: Cases of serogroup A meningococcal disease
- Community controls: Healthy members of the community controls matched with cases for age, sex and place of residence
- Hospital controls: Patients admitted to the hospital with an acute illness other than meningitis or septicemia

SUMMARY:
Major epidemics of meningococcal meningitis occur in countries of the African Sahel and sub-Sahel every few years. Most of these epidemics are caused by meningococci belonging to serogroup A. Until recently there has been no serogroup A conjugate vaccine available to prevent epidemics in Africa because none of the major pharmaceutical companies wanted to develop such a vaccine for commercial reasons. For this reason a public private partnership was established in 2001, the Meningitis Vaccine Project (MVP), with support from the Bill and Melinda Gates Foundation, to develop an affordable new serogroup A meningococcal conjugate vaccine for Africa. The new vaccine, MenAfriVac™, received WHO pre-qualification in 2010 and mass campaigns started in Burkina Faso, Mali and Niger in 2010. It is expected that full coverage through mass vaccination campaigns will be achieved by the end of 2011 in these three countries. A case-control study will be conducted in Mali and Niger during the epidemic seasons of 2012 and 2013 to assess the efficacy of MenAfriVac™.

DETAILED DESCRIPTION:
Massive epidemics of meningococcal disease continue to occur every few years in countries of the African Sahel and sub-Sahel - the African meningitis belt. In 2009 there were more than 50,000 reported cases in Nigeria alone. Most of these epidemics are caused by meningococci belonging to capsular polysaccharide serogroup A. African epidemics can be contained by existing meningococcal polysaccharide vaccines, saving many lives, but epidemics are not prevented by use of these vaccines. Recently, a new serogroup A meningococcal polysaccharide/protein conjugate vaccine (MenAfriVac), which may be able to prevent epidemics, was prequalified by the World Health Organization. This vaccine was developed by the Meningitis Vaccine Project (MVP) and is being produced at a cost ($0.40 per dose) that is affordable by countries of the African meningitis belt. Mass vaccination campaigns started in Burkina Faso, Mali and Niger at the end of 2010. Full coverage will be achieved in 2011 with progressive deployment to other countries in the meningitis belt.

The safety and immunogenicity of MenAfriVac have been established through phase 1 and phase 2 trials conducted in India and Africa but no efficacy trials have been undertaken. Prequalification was granted on the assumption that the high level of immunogenicity demonstrated in African populations would be reflected by a similar degree of efficacy. This is likely, but it is important that the efficacy of this vaccine is established definitively before large sums are spent on deploying the vaccine across the African meningitis belt. Therefore, a case control study to determine the efficacy of MenAfriVac in preventing serogroup A meningococcal meningitis in Mali and Niger is proposed.

A case-control study will be conducted in Mali and in Niger during the 2011, 2012 and 2013 meningitis seasons. Cases of meningitis will be detected through existing routine surveillance systems and their etiology established using standard microbiology or rapid diagnostic tests. Cases of proven serogroup A meningococcal meningitis (culture, antigen or PCR positive) will be matched with two hospital and two community controls who will, in turn, be matched with the cases for age and place of residence. A questionnaire will be administered to cases and controls which asks about previous meningococcal vaccination and other risk factors for meningococcal disease which might confound or modify assessment of the impact of vaccination with MenAfriVac. A blood sample will be collected for measurement of serogroup A meningococcal bactericidal and tetanus antibodies, as well as total immunoglobulin levels. Determination of vaccination status will be facilitated by the fact that vaccination cards will be issued to all recipients at the time of vaccination by the mass vaccination teams. Vaccine efficacy will be determined by comparing the odds of exposure to MenAfriVac in cases and controls.

ELIGIBILITY:
Inclusion Criteria:

- Cases: i)consent to participate; ii) Laboratory confirmed serogroup A meningococcal disease established by examination of the CSF (turbid CSF or a white cell > 10 per ul) and evidence of a serogroup A meningococcal infection established by (a) culture of serogroup A meningococci from the cerebrospinal fluid, blood or other normally sterile fluid, (b) a positive CSF latex test for serogroup A meningococcal antigen, (c) a positive serogroup A dipstick assay or (d) a positive CSF PCR for serogroup A meningococcal infection; iii) 1 to 29 years old.

iii) In target 1-29 year age group at the time of vaccination with MenAfriVac.

- Hospital controls: i)consent to participate; ii)patients admitted to the hospital with an acute illness other than meningitis, matched to cases for age and sex

-Community controls: i)consent to participate; ii)Healthy members of the community, matched to cases for age and sex

Exclusion Criteria:

* Case:

  i)Refusal to participate in the study; ii) infants<1 year old and adults>29 years old
* Hospital controls:

  i)Refusal to participate in the study; ii)Previous history of meningitis; iii) Presence of symptoms that could indicate meningitis
* Community controls:

  i)Refusal to participate in the study; ii)Previous history of meningitis; iii) Presence of symptoms that could indicate meningitis

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases: Patients with serogroup A meningococcal meningitis
  Hospital controls: Patients admitted to the same hospital/health facility as the case with an acute illness other than meningitis or septicemia.
  Community controls:Healthy individuals recruited from the same community as the case
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
serogroup A meningococci disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Brian Greenwood, MD, Principal Investigator — London School of Hygiene and Tropical Medicine; James Stuart, MD, Study Director — London School of Hygiene and Tropical Medicine
Locations (2):
- Center for Vaccine Development, Bamako, Bamako, Mali
- Centre de Recherche Médicale et Sanitaire, CERMES, Niamey, Niamey, Niger